CLINICAL TRIAL: NCT05325307
Title: Effect of Acupressure Applied Before Cystectomy on Preoperative Anxiety Level: Three Blind Randomized Controlled Studies
Brief Title: Effect of Acupressure Applied Before Cystectomy on Preoperative Anxiety Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Tugba CAM YANIK, PhD Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Mersin Univ
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2023-10

CONDITIONS: Anxiety; Hemodynamic Instability
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, three-arm randomized controlled clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In the study, a researcher (T.Ç.Y.) will determine the acupressure and placebo points to be applied to patients. However, the researcher (Z.Y.) who will apply acupressure and placebo acupressure be blinded without knowing whether these points are acupressure or placebo points. Participants will not know that they are in the acupressure or placebo group. When the research is completed, the data of the control and study groups (A or B) will be transferred to the computer environment by a researcher independent of the research, and the data will be analyzed by a statistician and the findings will be reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure Group (experimental) (Experimental): The experimental group will be given acupressure.
  Interventions: Other: Acupressure
- Placebo Acupressure Group (control) (Placebo Comparator): The placebo group will be given placebo acupressure
  Interventions: Other: Placebo acupressure

INTERVENTIONS:
Other: Acupressure — The experimental group will start with HT7 points and continue LI4 and EX-NH3 points. The application will be carried out by determining the priority order of the points with the draw. Attention will be paid to the intensity and duration of the pressure deemed appropriate. Since the individuals' responses will differ, the stiffness and pressure will be adjusted according to the individual's sensitivity not to cause tissue damage. Before starting the application, around the area to be pressed for 20-30 seconds will be gently rubbed with palm. With the gentle rubbing of the surrounding tissue, the tension and tissue sensitivity in warming, relaxing and preparatory will be reduced, and the tissue will be relieved. After, the point determined will be pressed manually for 2 minutes.
  Arms: Acupressure Group (experimental)
Other: Placebo acupressure — In the placebo acupressure group , the points 1.5 cm away from the HT7, LI4, and EX-NH3 points will be applied for an average of 15 minutes. Less pressure will be applied.
  Arms: Placebo Acupressure Group (control)

SUMMARY:
This randomized controlled study evaluates the effect of acupressure application on the anxiety level patients undergoing cystectomy surgery. The hypothesis of this study is that acupressure reduces anxiety levels and stabilizes hemodynamic parameters.

DETAILED DESCRIPTION:
In the study, 60 patients will randomly assigned to acupressure and placebo acupressure groups. To the acupressure group (n = 30), an average of 15 minutes will be applied to the HT7 (heart), LI4 (liver) and EX-NH3 (the point between the two eyes). In the placebo acupressure group (n = 30), the points 1.5 cm away from the HT7, LI4, and EX-NH3 points will be applied for an average of 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research (signing the Informed Consent Form),
* Conscious and cooperative
* Speaks and understands Turkish,
* 18-65 years old,
* Before surgery,
* Stable general condition,
* No sensitivity in the area where acupressure/placebo acupressure will be applied,
* 15 July 2022 - 15 July 2023 hospitalized in the urology clinic,
* No active COVID-19 infection,
* Patients without any psychiatric diagnosis will be included.

Exclusion Criteria:

* Those who do not agree to participate in the research (who do not sign the Informed Consent Form)
* Conscious and uncooperative,
* Not speaking or understanding Turkish,
* Not between the ages of 18-65,
* No surgical intervention planned,
* The planned emergency surgical intervention,
* Unstable general condition,
* Sensitivity in the area where acupressure/placebo acupressure will be applied,
* Active COVID-19 infection,
* 15 July 2022 - 15 July 2023 who did not stay in the urology clinic,
* Patients with current psychiatric diagnosis will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Anxiety evaluated using the State Anxiety Scale | Change from before implementation and immediately after, 20th minute after acupressure
  Scores ranging from 20 to 80 points are obtained in the scale. In the total score obtained from the scale in scoring the scale, 0-19 points indicate the absence of anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, and 60-79 points indicate severe anxiety level. Higher state anxiety scores indicate that anxiety level is also high

SECONDARY OUTCOMES:
Systolic blood pressure | Change from before implementation and immediately after, 20th minute after acupressure
  Systolic blood pressure (SBP), mmHg
Diastolic blood pressure | Change from before implementation and immediately after, 20th minute after acupressure
  Diastolic blood pressure (DBP), mmHg
Heart rate | Change from before implementation and immediately after, 20th minute after acupressure
  Beats per minute
Respiratory rate | Change from before implementation and immediately after, 20th minute after acupressure
  Lung breathing
Peripheral oxygen saturation | Change from before implementation and immediately after, 20th minute after acupressure
  %, percentage of oxygenated hemoglobin in peripheral arterial blood

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Altun Ugras, PhD, Study Director — Mersin University; Mualla Yılmaz, PhD, Principal Investigator — Mersin University; Zeliha Yaman, PhD, Principal Investigator — Mersin University; Naciye Balbay, graduate, Principal Investigator — Mersin University
Locations (1):
- Turkey, Mersin University,, Mersin, Turkey/Mersin,Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No